CLINICAL TRIAL: NCT04284189
Title: Aftercare of Childhood Cancer Survivors in Switzerland - the ACCS Switzerland Project
Brief Title: Aftercare of Childhood Cancer Survivors in Switzerland
Acronym: ACCS
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Collaborators: University Children's Hospital Basel (Other); Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Katrin Scheinemann, Division Head of Pediatric Oncology-Hematology, Kantonsspital Aarau
Other Study IDs: 2018-02304
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Childhood Cancer; Survivorship; Transition
Keywords: Childhood Cancer Survivor; Transition of follow-up care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transition model — Transition of follow-up care of childhood cancer survivors to adult care

SUMMARY:
The Aftercare of Childhood Cancer Survivors in Switzerland (ACCS) study is a multicenter cohort study designed to investigate transition of follow-up care from pediatric oncology to adult care in a prospective and longitudinal way. The investigators collect data on preferences and expectations for follow-up care and transition to adult care by questionnaires in adolescent and young adult survivors of childhood cancer.

DETAILED DESCRIPTION:
Background: Every year over 300 children and adolescents up to the age of 18 years are newly diagnosed with cancer in Switzerland. Survival after childhood cancer has increased substantially over the last decades and 10-year survival now exceeds 85%. This results in an increasing numbers of childhood cancer survivors - currently around 7,000 survivors in Switzerland. Due to cancer treatment or the cancer itself, a large part of the childhood cancer survivors suffers from late effects. Early diagnosis and intervention can reduce morbidity and mortality due to late effects. Therefore, regular follow-up care, even beyond childhood, is very important, but transition from pediatric to adult follow-up care is a critical point. In Switzerland there are very different aftercare and transition models, although it is unclear which aftercare strategy is the best and meets the needs of survivors. The Aftercare of Childhood Cancer Survivors (ACCS) study aims to fill this gap.

Objectives: The main objective of the ACCS study is to identify the current needs of adolescent and young adult long-term survivors in terms of follow-up care by comparing three different transition practices. The secondary objective is to assess survivors' knowledge on their diagnosis, therapy and follow-up examinations longitudinally.

Methods: ACCS is a multicenter questionnaire-based study, including survivors from three pediatric oncology centers in Switzerland. Eligible survivors who already transitioned to adult care at start of the study once receive a letter explaining the purpose of the study, the study information, the informed consent form, and the questionnaire. The questionnaire asks about cancer knowledge and additionally includes validated scales on cancer worry, self-management skills, ongoing care, and expectations. The survivors send the documents back by a prepaid envelope. Eligible survivors before transition to adult care at start of the study receive a letter explaining the purpose of the study, the study information and informed consent form, and the first questionnaire two to four weeks before the next scheduled follow-up visit. They can either send the documents back before the visit or bring them to the visit. The participants receive three month after the visit a short questionnaire to assess cancer knowledge. Three month after the follow-up visit after transition (15 month after last visit in pure pediatric setting), the participants receive the first comprehensive questionnaire again.

Rationale and significance: There are very different aftercare and transition models in Switzerland, although it is unclear which follow-up care strategy best meets the needs of survivors. The data collected within the ACCS study helps to define which transition and follow-up care strategies and related factors are favoured by adolescent and young adult survivors. Adaption of transition processes to the needs of survivors improve adherence to follow-up care of adult childhood cancer survivors. As late effects increase with increasing time from treatment, adult survivors of childhood cancer are at particular risk to develop late effects and it is important that they continue follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* 5-year survivor of childhood cancer
* Diagnosis according to ICCC3 I-XII; Langerhans cell histiocytosis (LCH), Hemophagocytic lymphohistiocytosis (HLH)
* Age at diagnosis <18 years
* Age at study ≥16 years
* At study start in follow-up care at one of the three pediatric oncology centers (group before transition) or transitioned not before 2014 (group after transition).
* Written informed consent

Exclusion Criteria:

* Treatment only by means of surgery and without increased risk of late effects (e.g. teratoma)
* <5 years after therapy of a relapse or palliative situation
* Severe cognitive impairment, which makes it impossible to complete the questionnaire independently
* Insufficient knowledge of the German language
* Informed consent form not signed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of childhood cancer survivors, who were diagnosed in three Swiss pediatric oncology centers at age <18 years and are ≥5-year from diagnosis and age ≥16 years at study inclusion. Additionally, survivors are at study start in follow-up care at one of the three pediatric oncology centers (group before transition) or have been transitioned to adult care not before 2014 (group after transition)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Cancer Worry as part of transition readiness | Change from baseline to 3 month and 15 month
  Assessment via validated "Cancer Worry Scale"
Self-management as part of transition readiness | Change from baseline to 3 month and 15 month
  Assessment via validated "Self-Management Skill Scale"
Evaluation of needs for ongoing care as part of transition readiness | Change from baseline to 3 month and 15 month
  Assessment via validated "Scale for ongoing Care"
Evaluation of expectation for transition as part of transition readiness | Change from baseline to 3 month and 15 month
  Assessment via validated "Expectation Scale"

SECONDARY OUTCOMES:
Survivors' cancer specific knowledge | Change from baseline to 3 month and 15 month
  Assessment via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Scheinemann, MD, Principal Investigator — Kantonsspital Aarau
Locations (3):
- Switzerland (3):
  - Division of Oncology - Hematology, Department of Pediatrics, Kantonsspital Aarau, Aarau
  - Division of Oncology/ Hematology, University Children's Hospital Basel, Basel
  - Division of Oncology/ Hematology, Department of Pediatrics, Kantonsspital Lucerne, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denzler S, Otth M, Scheinemann K. Aftercare of Childhood Cancer Survivors in Switzerland: Protocol for a Prospective Multicenter Observational Study. JMIR Res Protoc. 2020 Aug 26;9(8):e18898. doi: 10.2196/18898. PMID 32845247